CLINICAL TRIAL: NCT03415737
Title: Validity of the Turkish Version of the Profile Fitness Mapping Neck Questionnaire for Patients With Neck Pain
Status: Completed | Type: Observational
Sponsor: HATİCE ÇETİN (Other)
Responsible Party: Sponsor-Investigator, HATİCE ÇETİN, MSc, Pt, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: 776348
Record Dates: First submitted 2018-01-08; First posted 2018-01-30 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Pain; Neck Pain; Evaluations, Diagnostic Self; Assessment, Self
MeSH Terms: conditions — Pain; Neck Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Profile Fitness Mapping Neck Questionnaire

SUMMARY:
As patients improve on one parametric result, the results on the other parametric may worsen, but the total score may not be affected. For this reason, it would be useful to make measurements that evaluate all the parameters of the patients. Thus, it would be more advantageous to score both pain and symptoms separately, as well as activity limitations. Therefore, neck specific surveys are needed to meet this need.

For this reason, this study was planned to determine the validity of the questionnaire named "Profile Fitness Mapping Neck Questionnaire" in patients with neck pain.

DETAILED DESCRIPTION:
The translation of the original version of "Profile Fitness Mapping Neck Questionnaire" to Turkish will be translated by two independent professional translators. Afterwards, a person without a medical history and a native English speaker will be translated into English again. Once the translation stages are complete, the translators will be brought together to discuss the two versions of the questionnaire. Then the final state will be translated into the main language of the questionnaire and the compliance will be checked.

First of all, people who have been suffering from low back pain for at least six months will complete the "Profile Fitness Mapping NeckQuestionnaire", "Neck Disability Index", "SF-36 health related quality of life questionnaire" and "Visual Analog Scale".

Seven days after the questionnaire, the "Profile Fitness Mapping Neck Questionnaire" will be completed again.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain for more than six months during activity or rest
* Having a problem with the neck based on clinical examination and story

Exclusion Criteria:

* Having neurological problems
* Having vestibular or cerebellar problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neck pain
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Profile Fitness Mapping Neck Questionnaire | Change from Baseline Profile Fitness Mapping Neck Questionnaire score (functional limitation and symptom score) at 1 week.
  This questionnaire measures symptoms and functional limitations about neck pain.

SECONDARY OUTCOMES:
Neck Disability Index | All of the participants will assess at baseline with this index.
  This questionnaire evaluates disability related with neck pain.
SF-36 health related quality of life questionnaire | All of the participants will assess at baseline with this questionnaire.
  This questionnaire evaluates quality of life.
Visual Analog Scale | All of the participants will assess at baseline with this scale.
  This scale evaluates severity of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjorklund M, Hamberg J, Heiden M, Barnekow-Bergkvist M. The ProFitMap-neck--reliability and validity of a questionnaire for measuring symptoms and functional limitations in neck pain. Disabil Rehabil. 2012;34(13):1096-107. doi: 10.3109/09638288.2011.635747. Epub 2011 Dec 12. PMID 22149067